CLINICAL TRIAL: NCT06885281
Title: A Phase Ib/II, Open-label, Multi-center Study of ZL-1310 in Participants With Selected Solid Tumors
Brief Title: A Study of ZL-1310 in Participants With Selected Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Collaborators: Zai Lab (US) LLC (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-1310-002
Record Dates: First submitted 2025-02-24; First posted 2025-03-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): ZL-1310 as a single agent
  Interventions: Drug: ZL-1310

INTERVENTIONS:
Drug: ZL-1310 — drug ZL-1310

SUMMARY:
A Phase Ib/II, Open-label, Multi-center Study of ZL-1310 in Participants With Selected Solid Tumors

DETAILED DESCRIPTION:
This is an open-label, multiple-center, phase Ib/II study of ZL-1310 in selected solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Adult men and women ≥18 years of age
* Participants must have histologically confirmed, locally advanced or metastatic NECs, and must have experienced disease progression on or after platinum-based therapy
* Participants must be willing to undergo a tumor biopsy or must provide archived tumor tissue sample
* Participants must have at least one measurable target lesion as defined by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Participants with another known malignancy that is progressing or requires active treatment within the last 2 years
* Clinically active central nervous system (CNS) metastases
* Participants with leptomeningeal metastasis
* Participants who have received any ADC with a payload of topoisomerase I inhibitor (e.g., exatecan derivative)
* Treatment with any systemic anti-cancer treatment or other investigational products/device within 3 weeks before the first dose of study treatment
* Non-palliative radiotherapy within 2 weeks prior to first dose of study treatment or a history of radiation pneumonitis
* Major surgery within 4 weeks of the first dose of study treatment
* Hypersensitivity to any ingredient of the study treatment
* Out of range value (as defined in protocol) within 10 days prior to the first dose of study treatment
* Impaired cardiac function or clinically significant cardiac disease within the last 3 months before administration of the first dose of the study treatment
* Lung-specific intercurrent clinically significant illnesses and any autoimmune, connective tissue, or inflammatory disorders including but not limited to pneumonitis
* Has a history of (noninfectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening
* Pregnant or nursing (lactating) women
* Participants who have been on concomitant strong CYP3A or CYP2D6 inhibitors within 14 days or 5 half-lives before the first dose of study treatment, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse-Events in Phase Ib | up to 24 months
  Number of subjects with treatment-emergent adverse events (TEAEs)
Incidence of Serious Adverse Events in Phase Ib | up to 24 months
  Number of subjects with serious adverse events (SAEs)
Evaluate antitumor activity of ZL-1310 as a single agent in Phase II | up to 24 months
  Confirmed objective response rate (ORR) determined by blinded independent central review (BICR) in Phase II

SECONDARY OUTCOMES:
Evaluate preliminary antitumor activity of ZL-1310 as a single agent in Phase Ib | up to 24 months
  1. BICR-determined confirmed ORR in Phase Ib
  2. Investigator-determined confirmed ORR in Phase Ib
Evaluate preliminary antitumor activity of ZL-1310 as a single agent in Phase II | up to 24 months
  Investigator-determined confirmed ORR in Phase II
Incidence of Treatment Emergent Adverse-Events in Phase II | up to 24 months
  Number of subjects with treatment-emergent adverse events (TEAEs)
Incidence of Serious Adverse Events in Phase II | up to 24 months
  Number of subjects with serious adverse events (SAEs)
Pharmacokinetics (PK): Time to maximum concentration (Tmax) of Total Antibody in all phases | up to 24 months
  Time to maximum concentration (Tmax) is a pharmacokinetic parameter that refers to the time it takes for a drug or substance to reach its highest concentration in the bloodstream or a specific body compartment after administration
Pharmacokinetics (PK): maximum concentration (Cmax) of Total Antibody in all phases | up to 24 months
  Maximum concentration (Cmax) is a key pharmacokinetic parameter. It represents the highest concentration of a drug or substance that is achieved in the bloodstream or a specific biological fluid or tissue after administration
Pharmacokinetics (PK): area under the concentration-time curve (AUC) of Total Antibody in all phases | up to 24 months
  Area under the concentration-time curve (AUC) is a pharmacokinetic parameter that quantitatively describes the total exposure of a drug in the body over a specific period of time
Pharmacokinetics (PK): apparent clearance (CL) of Total Antibody in all phases | up to 24 months
  Apparent clearance (CL) is a pharmacokinetic parameter that describes the rate at which a drug is removed from the body relative to the drug's concentration in the bloodstream or a specific body fluid
Pharmacokinetics (PK): terminal elimination half-life (T1/2) of Total Antibody in all phases | up to 24 months
  Terminal elimination half-life (T1/2) is a pharmacokinetic parameter that characterizes the time it takes for the concentration of a drug in the body to decrease by half during the terminal phase of drug elimination
Pharmacokinetics (PK): time to maximum concentration (Tmax) of Unconjugated payloads in all phases | up to 24 months
  Time to maximum concentration (Tmax) is a pharmacokinetic parameter that refers to the time it takes for a drug or substance to reach its highest concentration in the bloodstream or a specific body compartment after administration
Pharmacokinetics (PK): maximum concentration (Cmax) of Unconjugated payloads in all phases | up to 24 months
  Maximum concentration (Cmax) is a key pharmacokinetic parameter. It represents the highest concentration of a drug or substance that is achieved in the bloodstream or a specific biological fluid or tissue after administration
Pharmacokinetics (PK): area under the concentration-time curve (AUC) of Unconjugated payloads in all phases | up to 24 months
  The area under the concentration - time curve (AUC) is a pharmacokinetic parameter that quantitatively describes the total exposure of a drug in the body over a specific period of time
Pharmacokinetics (PK): apparent clearance (CL) of Unconjugated payloads in all phases | up to 24 months
  Apparent clearance (CL) is a pharmacokinetic parameter that describes the rate at which a drug is removed from the body relative to the drug's concentration in the bloodstream or a specific body fluid
Pharmacokinetics (PK): terminal elimination half-life (T1/2) of unconjugated payloads in all phases | up to 24 months
  Terminal elimination half - life (T1/2) is a pharmacokinetic parameter that characterizes the time it takes for the concentration of a drug in the body to decrease by half during the terminal phase of drug elimination
Assess immunogenicity of ZL-1310 in all phases | up to 24 months
  Incidence of anti-drug antibodies (ADAs) to ZL-1310 in all phases
Evaluate stability and control of disease in all phases | up to 24 months
  BICR- and investigator-determined disease control rate (DCR) in all phases
Evaluate durability of response in all phases | up to 24 months
  BICR- and investigator-determined duration of response (DOR) in all phases
Evaluate progression-free survival (PFS) in all phases | up to 24 months
  BICR- and investigator-determined PFS in all phases
Evaluate survival in all phases | up to 24 months
  Overall survival (OS) in all phases

CONTACTS AND LOCATIONS:
Locations (16):
- United States (7):
  - Zai Lab Site 2001, San Francisco, California
  - Zai Lab Site 2002, New York, New York
  - Zai Lab Site 2024, Cleveland, Ohio
  - Zai Lab Site 2004, Philadelphia, Pennsylvania
  - Zai Lab Site 2003, Dallas, Texas
  - Zai Lab Site 2007, Houston, Texas
  - Zai Lab Site 2006, Fairfax, Virginia
- China (9):
  - Zai Lab Site 1002, Beijing, Beijing Municipality
  - Zai Lab Site 1013, Beijing, Beijing Municipality
  - Zai Lab Site 1009, Xiamen, Fujian
  - Zai Lab Site 1016, Guangzhou, Guangdong
  - Zai Lab Site 1004, Guangzhou, Guangdong
  - Zai Lab Site 1012, Harbin, Heilongjiang
  - Zai Lab Site 1006, Changsha, Hunan
  - Zai Lab Site 1008, Changchun, Jilin
  - Zai Lab Site 1001, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No